CLINICAL TRIAL: NCT05936996
Title: Prospective Clinical Registry Evaluating Contemporary MANTA Outcomes
Acronym: ACCESS MANTA
Status: Completed | Type: Observational
Sponsor: Essential Medical, Inc. (Industry)
Collaborators: Vascular Solutions LLC (Industry); Teleflex Medical Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: ST-3659
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Femoral Arteriotomy Closure
Keywords: MANTA; Arterial Closure Device; Large Bore Closure Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: MANTA Vascular Closure Device — The MANTA® Vascular Closure Device consists of a 14F or 18F MANTA® Closure Device, a 14F or 18F Sheath with Introducer, and an 8F Depth Locator. In the U.S. and Canada, the MANTA® Vascular Closure Device is indicated for closure of femoral arterial access sites while reducing time to hemostasis following the use of 10-20F devices or sheaths (12-25F OD) in endovascular catheterization procedures.

SUMMARY:
This is an observational study designed to evaluate the safety and clinical outcomes of the MANTA® Vascular Closure Device (VCD) (the MANTA® Device) in TAVR procedures. The study will enroll participants who are undergoing a TAVR procedure. The purpose of this study is to examine and collect data on outcomes of contemporary MANTA® large bore closure in standard of care (SOC) TAVR procedures with on-label use of the MANTA® device including appropriate patient selection and proper vascular access.

DETAILED DESCRIPTION:
In the U.S. and Canada, the MANTA® Vascular Closure Device is indicated for closure of femoral arterial access sites while reducing time to hemostasis following the use of 10-20F devices or sheaths (12-25F OD) in endovascular catheterization procedures. In Israel, the 14F MANTA® is indicated for closure of femoral arterial access sites following the use of 10-14F devices or sheaths (maximum OD/profile of 18F), and the 18F MANTA® device is indicated for closure of femoral arterial access sites following the use of 15-18F devices or sheaths (maximum OD/profile of 25F). The purpose of the study is to examine and collect data on outcomes of contemporary MANTA® large bore closure in standard of care (SOC) TAVR procedures with on-label use of the MANTA® device including appropriate patient selection and proper vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Candidate meets criteria for on-label use of MANTA® VCD as specified in the country-specific MANTA® VCD Instructions for Use (IFU), per judgement of the investigator.
* Age ≥21 years

Exclusion Criteria:

* Unable or unwilling to give informed consent or unwilling to complete follow-up assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Qualifying subjects undergoing TAVR using the MANTA® VCD for large bore closure.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of VARC-3 Major & Minor Vascular complications | within 30 days of TAVR procedure
Time to Hemostasis | During the procedure
  The elapsed time between MANTA® deployment and first observed and confirmed arterial hemostasis

SECONDARY OUTCOMES:
Additional interventions: Required at large bore access site to address complications | within 30 days following the procedure
  The percentage of subjects with additional interventions required at large bore access site to address bleeding or other large bore access site complications (e.g., bare or covered stent or surgical repair), within 30 days following the procedure
Technical Success: | During the procedure
  The percentage of subjects in whom closure is obtained with the MANTA® VCD without the use of unplanned endovascular or surgical intervention
Ambulation Success: | During procedure admission
  The percentage of a previously ambulatory subjects (until day of TAVI) who are able to ambulate for at least 20 feet/6 meters without re-bleeding.
Treatment Success: | within 30 days of TAVR procedure
  The percentage of subjects in whom the time to Hemostasis ≤10 minutes and have no Large Bore Access Related Major VARC-3 complications within 30 days.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Baptist Health Medical Center-Jacksonville, Jacksonville, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Henry Ford Health, Detroit, Michigan
  - University at Buffalo, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White - Round Rock, Round Rock, Texas
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data obtained will be used, without mentioning Subject PHI, to assess the results of the research, and the data could be used in the future with regard to this study or other studies. The data can be passed on to the health authorities for the purposes of registering the medical device.